CLINICAL TRIAL: NCT03031964
Title: Survivorship, Clinical and Functional Outcomes of the Multihole Revision Acetabular Cup
Brief Title: Survivorship, Radiographic, and Functional Outcomes of the Multihole Revision Acetabular Cup
Status: Terminated | Type: Observational
Why Stopped: Closed the single investigator initiated study at request of Stryker, to begin collecting as a multicenter study.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Staff Surgeon, The Cleveland Clinic
Other Study IDs: #16-1030
Record Dates: First submitted 2016-12-20; First posted 2017-01-26 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Complications Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- revision multihole acetabular cup: Revision total hip arthroplasty using multihole revision acetabular cup
  Interventions: Device: revision multihole acetabular cup

INTERVENTIONS:
Device: revision multihole acetabular cup — post market study of multi hole revision acetabular cup
  Other Names: Stryker restoration anatomic shell

SUMMARY:
This study will evaluate patients receiving a multihole revision acetabular implant for total hip arthroplasty (THA) and will be followed for 10 years to collect data on survivorship of the implanted prosthesis.

DETAILED DESCRIPTION:
Data will be collected preoperatively, and at the standard of care (SOC) office visits at 4 weeks, 1 year, 2 years, 5 years and 10 years postoperatively. The research coordinator at each site will identify, recruit, and prospectively follow the 60 patients at his/her site. Patient demographics (e.g., age, gender, body mass index (BMI)), comorbidities, reason for revision, Paprosky classification, native femoral head measurement (mm) etc. will be collected preoperatively. The study coordinator will contact patients prior to each visit to ensure patient compliance. At each visit, A-P and cross-lateral radiographic evaluation (i.e., use of Engh classification to quantify osteolysis/loosening) will occur. In addition, patients will be assessed for any complications (e.g., dislocation, emergency department visits, infection, reoperation, etc.). Patients will complete the Hip disability and Osteoarthritis Outcome Score (HOOS) and Veterans Rand 12 (VR-12) forms (including a specific question regarding groin pain) and a pain assessment. In the event that a patient has relocated and/or refuses to return to the office for the 5-year visit, a script will be sent to the patient to have x-rays done and sent to the PI, and questionnaires will be mailed. All data will be entered and maintained in RedCap.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring revision total hip replacement of the acetabular component or complicated primary total hip replacement.
2. Femoral stem (either retained or replaced) is a compatible Stryker stem.
3. Patient is willing to comply with follow-up requirements (e.g. will return for long-term follow-up visits)
4. Age: 18-85 years

Exclusion Criteria:

1. Patient has a BMI > 40
2. Exclude revision for infection
3. Patient is undergoing bilateral THA surgery or had prior hip arthroplasty on contralateral side less than 6 months from date of surgery
4. Patient has history of radiation therapy
5. Patient has known diagnosis of renal disease
6. Patient has known diagnosis of osteoporosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a revision total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-12; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
survivorship of a multihole revision acetabular cup | 10 years
  evaluate standard of care radiographs for any signs of implant compromise such as loosening or osteolysis

SECONDARY OUTCOMES:
Clinical outcomes of multihole revision acetabular cup | 10 years
  determine clinical outcomes with VR-12 surveys
functional outcomes of multihole revision acetabular cup | 10 years
  determine functional outcomes with HOOS surveys
assess pain levels in patients who receive multihole revision acetabular cup | 10 years
  determine level of pain with pain assessments

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Higuera, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jafari SM, Bender B, Coyle C, Parvizi J, Sharkey PF, Hozack WJ. Do tantalum and titanium cups show similar results in revision hip arthroplasty? Clin Orthop Relat Res. 2010 Feb;468(2):459-65. doi: 10.1007/s11999-009-1090-5. PMID 19809857
- [Background] Kremers HM, Howard JL, Loechler Y, Schleck CD, Harmsen WS, Berry DJ, Cabanela ME, Hanssen AD, Pagnano MW, Trousdale RT, Lewallen DG. Comparative long-term survivorship of uncemented acetabular components in revision total hip arthroplasty. J Bone Joint Surg Am. 2012 Jun 20;94(12):e82. doi: 10.2106/JBJS.K.00549. PMID 22717834
- [Background] Unger AS, Lewis RJ, Gruen T. Evaluation of a porous tantalum uncemented acetabular cup in revision total hip arthroplasty: clinical and radiological results of 60 hips. J Arthroplasty. 2005 Dec;20(8):1002-9. doi: 10.1016/j.arth.2005.01.023. PMID 16376255
- [Background] Odri GA, Padiolleau GB, Gouin FT. Oversized cups as a major risk factor of postoperative pain after total hip arthroplasty. J Arthroplasty. 2014 Apr;29(4):753-6. doi: 10.1016/j.arth.2013.07.001. Epub 2013 Aug 6. PMID 23927907
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Silverton CD, Rosenberg AG, Sheinkop MB, Kull LR, Galante JO. Revision total hip arthroplasty using a cementless acetabular component. Technique and results. Clin Orthop Relat Res. 1995 Oct;(319):201-8. PMID 7554631
- [Background] Petrera P, Rubash HE. Revision Total Hip Arthroplasty: The Acetabular Component. J Am Acad Orthop Surg. 1995 Jan;3(1):15-21. doi: 10.5435/00124635-199501000-00003. PMID 10790649
- [Background] Klika AK, Murray TG, Darwiche H, Barsoum WK. Options for acetabular fixation surfaces. J Long Term Eff Med Implants. 2007;17(3):187-92. doi: 10.1615/jlongtermeffmedimplants.v17.i3.20. PMID 19023943
- [Background] Ramappa M, Bajwa A, Kulkarni A, McMurtry I, Port A. Early results of a new highly porous modular acetabular cup in revision arthroplasty. Hip Int. 2009 Jul-Sep;19(3):239-44. doi: 10.1177/112070000901900309. PMID 19876878
- [Background] Frenkel SR, Jaffe WL, Dimaano F, Iesaka K, Hua T. Bone response to a novel highly porous surface in a canine implantable chamber. J Biomed Mater Res B Appl Biomater. 2004 Nov 15;71(2):387-91. doi: 10.1002/jbm.b.30104. PMID 15389510
- [Background] Paprosky WG, Perona PG, Lawrence JM. Acetabular defect classification and surgical reconstruction in revision arthroplasty. A 6-year follow-up evaluation. J Arthroplasty. 1994 Feb;9(1):33-44. doi: 10.1016/0883-5403(94)90135-x. PMID 8163974
- [Background] Claus AM, Engh CA Jr, Sychterz CJ, Xenos JS, Orishimo KF, Engh CA Sr. Radiographic definition of pelvic osteolysis following total hip arthroplasty. J Bone Joint Surg Am. 2003 Aug;85(8):1519-26. doi: 10.2106/00004623-200308000-00013. PMID 12925632